CLINICAL TRIAL: NCT02323178
Title: A Phase I/II Study of Eltrombopag in Patients With Chronic Myelomonocytic Leukemia and Thrombocytopenia
Brief Title: A Study of Eltrombopag in Patients With CMML and Thrombocytopenia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Collaborators: GlaxoSmithKline (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFM-LMMC-Eltrombopag; 2013-001779-19 (EudraCT Number)
Record Dates: First submitted 2014-05-26; First posted 2014-12-23 (Estimated); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: CMML; Thrombocytopenia
Keywords: Chronic myelomonocytic leukemia; thrombocytopenia; eltrombopag
MeSH Terms: conditions — Thrombocytopenia; Leukemia, Myelomonocytic, Chronic | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- eltrombopag (Experimental)
  Interventions: Drug: eltrombopag

INTERVENTIONS:
Drug: eltrombopag — initial dose of 50 mg once daily, then the dose can be sequentially increased every 2 weeks up to a maximum dose of 300mg/day
  Other Names: revolade

SUMMARY:
Treatment of patients with chronic myelomonocytic leukemia (CMML) and thrombocytopenia.

DETAILED DESCRIPTION:
All eligible patients will be treated with eltrombopag for a minimum of twelve weeks and a maximum of 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Chronic myelomonocytic leukemia (CMML) according to WHO criteria:
* Stable excess in blood monocytes > 1 G/L
* Lack of bcr-abl rearrangement (or Philadelphia chromosome)
* Bone marrow blast cells < 20%
* Dysplasia of at least one lineage or clonality marker or blood monocytosis during more than 3 months w/o other explanation
* Platelet counts < 50 G/L on two successive blood counts in the 2 weeks preceding inclusion
* Either of D1 or D2 criteria:
* Lack of features of advanced disease If white blood cell count (WBC) < 13 G/L: International Prognostic Scoring System (IPSS) low or intermediate-1

If WBC ≥ 13 G/L: no more than one of the following criteria:

* Clonal cytogenetic abnormality other than t(5;12) (q33; p13)
* Absolute neutrophil count (ANC) > 16 G/L
* Anemia (Hb < 100 g/L)
* Extramedullary localization (documented cutaneous, pleural or pericardial effusion, etc…) OR D2- Features of advanced disease If WBC < 13 G/L: IPSS intermediate-2 or high

If WBC ≥ 13 G/L: two or more of the following criteria:

* Clonal cytogenetic abnormality other than t(5;12) (q33; p13)
* ANC > 16 G/L
* Anemia (Hb < 100 g/L)
* Extramedullary localization (documented cutaneous, pleural or pericardial effusion, etc…) And having resisted (progression or stable disease without hematological improvement according to International Working Group (IWG) 2006 criteria) or relapsed after a treatment with a hypomethylating agent (azacitidine or decitabine for a minimum of 6 cycles)
* Blast cells ≤ 5% in the bone marrow
* Performance status 0-2 on the Eastern Cooperative Oncology Group (ECOG) Scale
* Serum Creatinin < 2 times the upper limit of normal (ULN)
* Alanine transaminase (ALT) and aspartate transaminase (AST) < 3 ULN, total bilirubin < 1.5 ULN (except Gilbert Syndrome)
* Adequate contraception if relevant
* Signed informed consent

Exclusion Criteria:

* CMML with t(5 ;12) or Platelet-derived growth factor beta receptor (PDGFbetaR) rearrangement
* Acute blastic transformation of CMML with bone marrow blast cells > 20%
* Bone marrow blast cells > 5%
* Patients eligible for allogeneic bone marrow transplantation with an identified donor
* Intensive chemotherapy given less than 3 months before inclusion
* Pregnant or breastfeeding
* Hepatitis C infection
* Splenomegaly > 16 cm by ultrasound or CT scan (Not Applicable in patients without palpable splenomegaly)
* Significant (grade II-IV) myelofibrosis (bone marrow trephine if bone marrow aspirate with poor cellularity, or features of myelofibrosis on the peripheral blood smear (teardrop erythrocytes)
* Clinically relevant thromboembolic risk factor which, in the investigator's opinion, is such that the benefit/risk ratio becomes unfavourable if platelet counts increase
* Liver cirrhosis (Child-Pugh score ≥ 5)
* Prior Cancer (except in situ cervix carcinoma, limited basal cell carcinoma, or other tumors if not active during the last 3 years)
* Serious concomitant systemic disorder, including active bacterial, fungal or viral infection that, in the opinion of the investigator, would compromise the safety of the patient and/or his/her ability to complete the study.
* Hypersensitivity to Eltrombopag

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-08-07 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Platelet response | 12 weeks
  Hematological improvement after twelve weeks of eltrombopag treatment

SECONDARY OUTCOMES:
Duration of platelet response | 30 months
  Duration of platelet response at end of follow-up

OTHER OUTCOMES:
safety of eltrombopag assessed by clinical and biological toxicity of eltrombopag evaluated using NCI CTCAE v4.0 | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël Itzykson, MD, Principal Investigator — Saint-Louis Hospital, Paris, France; Pierre Fenaux, MD, PHD, Study Director — Saint-Louis Hospital, Paris, France
Locations (26):
- France (26):
  - CHU d'Amiens, Amiens
  - CHU d'Angers, Angers
  - CH Victor Dupouy, Argenteuil
  - Hôpital Avicenne, Bobigny
  - Hôpital privé Sévigné, Cesson-Sévigné
  - CHU Henri Mondor, Créteil
  - CHU de Grenoble, Grenoble
  - CH Le Mans, Le Mans
  - CHRU de Limoges, Limoges
  - Centre Hospitalier Lyon Sud, Lyon
  - Institut Paoli Calmettes, Marseille
  - Centre Hospitalier de Meaux, Meaux
  - CHU de Nantes, Nantes
  - Centre Catherine de Sienne, Nantes
  - Hôpital Archet 1, Nice
  - Hôpital Saint Louis - Service d'hématologie AJA, Paris
  - Hôpital Saint Louis - Service d'hématologie séniors, Paris
  - CHU de Haut-Lévèque, Pessac
  - CHU de Poitiers, Poitiers
  - Centre Hospitalier de la région d'Annecy, Pringy
  - Hôpital Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - IUCT Oncopole - Médecine interne, Toulouse
  - IUCT Oncopole - Service d'Hématologie Clinique, Toulouse
  - CHU Brabois, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif